CLINICAL TRIAL: NCT03473574
Title: A Randomized Phase II Trial of Durvalumab and Tremelimumab With Gemcitabine or Gemcitabine and Cisplatin Compared to Gemcitabine and Cisplatin in Treatment-naïve Patients With Cholangio- and Gallbladder Carcinoma (IMMUCHEC)
Brief Title: Durvalumab and Tremelimumab With Gemcitabine or Gemcitabine/Cisplatin Compared to Gemcitabine/Cisplatin in CCA Patients
Acronym: IMMUCHEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-HEP-0117; 2017-001538-25 (EudraCT Number)
Record Dates: First submitted 2018-03-14; First posted 2018-03-22 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Cholangiocarcinoma; Gall Bladder Carcinoma; Cholangiocarcinoma Non-resectable; Gallbladder Carcinoma Non-Resectable
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms | interventions — durvalumab; Gemcitabine; Cisplatin; tremelimumab

STUDY DESIGN:
Intervention Model Description: Treatment Arm A: Combination of Durvalumab, Tremelimumab (Regimen 1) and Gemcitabine Treatment Arm B: Combination of Durvalumab, Tremelimumab (Regimen 1), Gemcitabine and Cisplatin Treatment Arm C: Gemcitabine and Cisplatin Treatment Arm D: Combination of Durvalumab, Tremelimumab (Regimen 2), Gemcitabine and Cisplatin Treatment Arm E: Combination of Durvalumab, Gemcitabine and Cisplatin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm A (Experimental): Durvalumab in combination with Tremelimumab (Regimen 1) and Gemcitabine
  Interventions: Biological: Durvalumab; Drug: Gemcitabine; Biological: Tremelimumab
- Arm B (Experimental): Durvalumab in combination with Tremelimumab (Regimen 1), Gemcitabine and Cisplatin
  Interventions: Biological: Durvalumab; Drug: Gemcitabine; Drug: Cisplatin; Biological: Tremelimumab
- Arm C (Other): Gemcitabine in combination with Cisplatin
  Interventions: Drug: Gemcitabine; Drug: Cisplatin
- Arm D (Experimental): Durvalumab in combination with Tremelimumab (Regimen 2), Gemcitabine and Cisplatin
  Interventions: Biological: Durvalumab; Drug: Gemcitabine; Drug: Cisplatin; Biological: Tremelimumab
- Arm E (Experimental): Durvalumab in combination with Gemcitabine and Cisplatin
  Interventions: Biological: Durvalumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Biological: Durvalumab — immune checkpoint inhibitor
  Arms: Arm A; Arm B; Arm D; Arm E
Drug: Gemcitabine — standard chemotherapy
Drug: Cisplatin — standard chemotherapy
  Arms: Arm B; Arm C; Arm D; Arm E
Biological: Tremelimumab — immune checkpoint inhibitor
  Arms: Arm A; Arm B; Arm D

SUMMARY:
To determine the efficacy in terms of objective response rate (ORR) of the combination of durvalumab and tremelimumab in addition with gemcitabine or in addition with gemcitabine and cisplatin in treatment-naïve patients with advanced, unresectable and/or metastatic cholangio- and gallbladder carcinoma (CCA).

DETAILED DESCRIPTION:
Patients with CCA have poor outcomes, as a consequence of the very aggressive nature of the disease, and the limited treatment options. Thus there is a significant unmet medical need for additional treatment options for use in this patient population. As in most other tumor entities however, only a fraction of patients respond to immunotherapy alone. Evidence suggests that those patients might preferentially have tumors that have favorable mutational landscapes, express the PD-L1 and/ or contain preexisting tumor-infiltrating CD8+ T cells that are inhibited locally, e.g., by PD-1 engagement. In order to increase the proportion of patients who could ultimately benefit from immunotherapies, it is important to develop strategies that can be employed for converting tumor microenvironments lacking T cell infiltration to ones displaying antitumor T-cell immunity and therefore to sensitize tumors to checkpoint inhibition therapy. Therefore, the aim of this study is to determine the combination of durvalumab and tremelimumab in addition with gemcitabine or in addition with gemcitabine and cisplatin in treatment-naïve patients with advanced, unresectable and/or metastatic cholangio- and gallbladder carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Fully-informed written consent and locally required authorization (European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Age ≥ 18 years.
3. Histologically documented diagnosis of cholangiocarcinoma or gall bladder carcinoma and available tumor tissue (block or at least 4 slides) for translational research.
4. Performance status (PS) ≤ 1(ECOG scale).
5. At least one measurable site of disease as defined by RECISTv1.1 criteria.
6. Adequate bone marrow and renal function including the following: Hemoglobin

   ≥ 9.0 g/dL; absolute neutrophil count ≥ 1.5 x 10^9/L; platelets ≥ 100 x 10^9 /L; Creatinine ≤ 1.5 x upper normal limit.
7. Calculated creatinine clearance ≥40 mL/min as determined by the Cockcroft- Gault equation (using actual body weight)
8. Adequate hepatic function (with stenting for any obstruction, if required) including the following: Total bilirubin ≤ 2x upper normal limit; AST (SGOT), ALT (SGPT) ≤ 5 x upper normal limit; prothrombin time ≥ 60%; albumin ≥ 30 g/L.
9. Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.
10. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered postmenopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
11. The patient is willing and able to comply with the protocol for the duration of the study, including hospital visits for treatment and scheduled follow-up visits and examinations.

Exclusion Criteria:

1. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study, or during the follow-up period of an interventional study
2. Participation in another clinical study with an investigational product within 21 days prior to the first dose of the study treatment.
3. Prior immunotherapy or use of other investigational agents, including prior treatment with an anti-Programmed Death receptor-1 (PD-1), anti-Programmed Death-1 ligand-1 (PD-L1), anti-PD-L2, or anti-cytotoxic T-lymphocyte associated antigen-4 (anti-CTLA-4) antibody, therapeutic cancer vaccines.
4. Prior chemotherapy with gemcitabine, Cisplatin and/or capecitabine (exception: gemcitabine, cisplatind and/or capecitabine in the adjuvant setting, last infusion has to be ≥ 6 months prior randomization).
5. Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
6. Any concurrent chemotherapy, IMP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable. Note: Local treatment of isolated lesions for palliative intent is acceptable (eg, local radiotherapy).
7. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drugs.
8. Major surgery (as defined by the Investigator) within 4 weeks prior to the first dose of the investigational product (IMP) of starting the study and patients must have recovered from effects of major surgery. Note: Local non-major surgery for palliative intent (eg, surgery of isolated lesions, per-cutaneous biliary drainage or biliary stenting) is acceptable.
9. History of allogenic organ transplantation.
10. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], celiac disease, systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]).

    The following are exceptions to this criterion:
    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
11. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
12. History of another primary malignancy except for:

    * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IMP and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
13. History of leptomeningeal carcinomatosis
14. Brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have a CT/ MRI of the brain prior to study entry.
15. History of active primary immunodeficiency
16. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen [HBsAg) result], hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
17. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication) Receipt of live attenuated vaccine within 30 days prior to the first dose of IMP.

Note: Patients, if enrolled, should not receive live vaccine whilst receiving IMP and up to 30 days after the last dose of IMP. 19. Body weight ≤30 kg. 20. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of tremelimumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy. 21. Known allergy or hypersensitivity to any of the IMPs or any of the constituents of the product. 22. Prior randomisation or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment. 23. Any co-existing medical condition that in the investigator's judgement will substantially increase the risk associated with the patient's participation in the study. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG. 25. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 30 months
  Response Rate (RR) according to RECIST V1.1

SECONDARY OUTCOMES:
Overall survival (OS) | max observation period 30 months
  Efficacy of the combination of durvalumab and tremelimumab in addition with gemcitabine or in addition with gemcitabine and cisplatin in treatment naïve patients with advanced, unresectable and/or metastatic cholangio- and gallbladder carcinoma
Incidence of Treatment Emergent Adverse Events as assessed by NCI CTCAE V4.0 (Safety and Tolerability) | 30 months
  Data will be obtained on vital signs, clinical parameters and feasibility of the regimen
Quality of Life | 30 months
  EORTC-QLQ-C30 (European Organisation for Research and Treatment of Cancer - Quality of Life Core Questionnaire 30 items) Version 3.0. The QLQ-C30 is composed of multi-item scales and single-item measures, including fiveAll of the scales and single-item measures have a score range from 0 to 100. A high score shows a high response level. A high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems functional scales, three symptom scales, a global health status / QoL scale, and six single items.

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Vogel, Prof. Dr., Principal Investigator — Hannover Medical School
Locations (1):
- Medizinische Hochschule Hannover, Klinik für Gastroenterologie, Hepatologie & Endokrinologie, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: AIO - Working Group for Medical Oncology from the German Cancer Society — http://www.aio-portal.de/
- See also: Description AIO-Studien-gGmbH — http://www.aio-portal.de/